CLINICAL TRIAL: NCT05138588
Title: Personalized Repetitive Transcranial Magnetic Stimulation (rTMS) in Cognitive Fluctuations of Dementia With Lewy Bodies (DLB): Proof of Concept
Acronym: STIMLEWY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8238
Record Dates: First submitted 2021-11-02; First posted 2021-12-01 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Dementia With Lewy Bodies Diagnosis; Significant Cognitive Fluctuations in DLB
Keywords: rTMS; arousal; DLB; fluctuations; insula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All investigators, participants, care providers and outcome assessors will be blinded, with the exception of the investigator programming the stimulation sequences and the nurses administrating the rTMS sequences.
  For the investigators, the unblinding and the taking of knowledge of the subjects in each group will take place after the end of any experimental run, during the data processing phase. In the event of serious adverse events, the unblinding will be carried out before the end of the research.
  For participants, the unblinding will take place at the end of the last follow-up visit of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VERUM (Experimental): In the "verum" experimental condition, participants will receive the experimental rTMS stimulation sessions, meaning the rTMS sessions targeting the insular cortex, taking into account the insular hypoperfusion (through MRI images) of each patient.
  Interventions: Device: rTMS
- CONTROL (Sham Comparator): In the "control" experimental condition, participants will receive the control rTMS stimulation sessions, meaning the rTMS sessions will target the occipital cortex.
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — For each subject, a verum condition and a control condition will be programmed. We will use the QPS-5 method (4 pulses, Inter-Stimulation Interval; ISI: 5 seconds).
  Other Names: Repetitive Magnetic Transcranial Stimulation is a non-invasive neuromodulation technique based on the principle of electromagnetic induction.

SUMMARY:
The present study is a monocentric, therapeutic clinical trial involving forty patients diagnosed with Dementia with Lewy Bodies (DLB). The aim of this clinical trial is to evaluate the feasibility and relevance of repetitive transcranial magnetic stimulation (rTMS); a non-invasive neuromodulation technique, with a main emphasis on the evaluation of the outcome on cognitive fluctuations. For this purpose, we will compare two distinct rTMS conditions (control and experimental) in a pre-post rTMS setting. The experimental condition will be targeting the insular cortex which has been shown to be affected at prodromal DLB stages, in the form of decreased grey matter concentration and a decreased regional Cerebral Blood Flow (rCBF hypoperfusion) [Blanc et al., 2015 ; Roquet et al., 2016 ; Roquet et al., 2017]. Furthermore, these insular alterations are correlated to cognitive fluctuations [Chabran et al., 2020]. In DLB, cognitive fluctuations are particularly pervasive and manifest in the form of alertness alterations and modifications of arousal states. Participants will repeatedly undergo a series of clinical and cognitive assessments in addition to several neuroimaging examinations, namely multimodal Magnetic Resonance Imaging (MRI) and electroencephalogram (EEG) recordings, in order to evaluate potential physiological modifications and clinical changes of symptoms, pre-/post-rTMS.

DETAILED DESCRIPTION:
Objectives:

* To provide a proof of concept by validating the hypoactivity (hypoperfusion) of the anterior insula ("AI biomarker") as a causal factor of the instability of arousal states in DLB.
* To evaluate if improvement of arousal translates clinically into a reduction of cognitive fluctuations and an improvement of other functional parameters (clinical measures of symptoms).
* Evaluation of the relevance of the AI biomarker as a predictive tool for clinical response.
* Assessment of reproducibility of the AI hypoperfusion (biomarker) at an individual level and thereby its potential as a diagnostic or therapeutic biomarker.
* Collection, description and analysis of all adverse events and required information for the implementation of future phase II and III studies

Methodological approach:

The present study will be conducted at the "non-invasive neurostimulation center of Strasburg" (Centre de Neuromodulation Non-invasive de Strasbourg ; CEMNIS) in collaboration with the Memory Clinic of Strasbourg (Centre Mémoire de Ressources et de Recherches ; CM2R) of the University Hospitals of Strasbourg (HUS) and the ICube laboratory (Team IMIS, UMR 7357, CNRS). We propose a single-centre, two-arm, randomized, crossover, double-blind comparative study. N=40 patients will be prospectively recruited in order to create two experimental groups (arms) (Group A and Group B) in a cross-over study design, following two experimental phases (I and II). The protocol will include two rTMS conditions: (1) verum stimulation (target: insular cortex) and (2) control stimulation (target: occipital cortex). The running order for each participant will be counterbalanced: Group A will start with the verum rTMS in phase I, followed by the control rTMS in phase II. Group B will start with the control rTMS in phase I, followed by the verum rTMS in phase II. One phase of rTMS will consist of a total of ten visits. One visit will include two sessions of rTMS, summing up to a total of twenty sessions of rTMS for each patient. Participants will undergo multiple EEG recordings and multimodal cerebral MRI scans, as well as several different clinical assessments (self-reported, reported by the investigator and the patients' main caregiver) numerous times during the protocol, pre- and post-rTMS sessions. In sum, each patient will undergo five MRI scans and three clinical assessments. The clinical trial schedules a total of N=37 visits for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient aged ≥ 45 years
* Enrolled in a social health insurance scheme
* Diagnosed with probable DLB according to McKeith et al. criteria, 2017, or McKeith et al. 2020 criteria for the prodromal stage
* A Mini Mental State Examination (MMSE; Folstein et al., 1983) score ≥ to 18 in the last 6 months (prodromal stage or a major neurocognitive disorder (dementia syndrome) at moderate stage)
* MMSE score ≥ to 15 at the inclusion visit
* Presence of clinically significant cognitive fluctuations
* Caregivers of eligible patients do have to be able to stay with the patient for at least 4 hours a day, 3 days a week, and have to be able to provide requested information and accompany the patient to the certain visits.
* The patient must be able to understand the objectives and risks of the study and has to be able to give dated and signed informed consent. In the case of a designed guardian or curator, the guardian or curator will sign the consent.
* For women of childbearing age, effective contraception throughout the study is required

Exclusion criteria:

* History of generalized seizures (epilepsy)
* Pharmacological treatment for cognitive fluctuations in DLB with dose modifications that have taken place less than 2 months before the first visit of the protocol (anticholinesterase and neuroleptics)
* Anti-epileptic drug treatment "Keppra" (Levetiracetam)
* History of psychosis or severe depression unrelated to DLB
* History of brain surgery (tumour removal, electrode implantation, certain strokes as judged by the investigator, oedema...)
* Patients with any contraindication for MRI scans (claustrophobia, pacemaker, cochlear implant, mechanical heart valve, metallic prostheses, neurostimulators, other non-removably implanted electronic medical devices etc.)
* Subject unable to understand the aims and risks of the study and patients unable to give full informed consent
* Having a MMSE score < to 18 in the last 6 months (prodromal stage or mild to moderate dementia)
* MMSE score < to 15 at the inclusion visit
* Patients in an emergency or life-threatening situation
* Patients under court protection
* Pregnancy
* Breastfeeding
* Patients in exclusion period (determined by a previous or current study)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Electroencephalogram measures | Primary outcome measures will be realized one week before each rTMS stimulation phase.
  The primary endpoint will be the comparison of the intensity of fluctuations in arousal level
Electroencephalogram measures | Primary outcome measures will be realized one week after each rTMS stimulation phase.
  The primary endpoint will be the comparison of the intensity of fluctuations in arousal level

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric BLANC, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No